CLINICAL TRIAL: NCT02104258
Title: Rehabilitation of Acute Hamstring Injuries in Male Athletes: A Prospective Single-site Randomized Controlled Clinical Trial Comparing Two Rehabilitation Protocols With Different Emphasis on Eccentric Exercises
Brief Title: Rehabilitation of Acute Hamstring Injuries in Male Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspetar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HAR47; CMO/000047/fj (Other: Aspetar)
Record Dates: First submitted 2014-03-22; First posted 2014-04-04 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Strains
Keywords: Hamstring; Muscle; Injury; Treatment; Rehabilitation
MeSH Terms: conditions — Sprains and Strains; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy ASPETAR (Active Comparator): The patients will follow the ASPETAR Hamstring Rehabilitation Protocol, which is a standardised physiotherapy protocol, including range of motion exercises, progressive strengthening exercises, core stability training and agility exercises [10].
  The ASPETAR protocol consist of predefined rehabilitation stages including sports specific stages. Specific functional based criteria for progression will be utilized for each of the six rehabilitation stages. No pain provocation when performing the exercises will be allowed.
  The rehabilitation will be initiated as soon as possible after inclusion and the patients will be supervised by experienced physiotherapists in the Rehabilitation Department at Aspetar 3 to 5 days per week.
  Interventions: Other: Physiotherapy ASPETAR
- Physiotherapy ASPETAR+ (Active Comparator): The patients will follow the ASPETAR+ Hamstring Rehabilitation Protocol. ASPETAR+ is similar to ASPETAR, but consists of additional lengthening exercises which will be initiated early in the rehabilitation phase.
  ASPETAR+ consist of predefined rehabilitation stages including sports specific stages. Specific functional based criteria for progression will be utilized for each of the six rehabilitation stages. No pain provocation when performing the exercises will be allowed.
  The rehabilitation will be initiated as soon as possible after inclusion and the patients will be supervised by experienced physiotherapists in the Rehabilitation Department at Aspetar 3 to 5 days per week.
  Interventions: Other: Physiotherapy ASPETAR+

INTERVENTIONS:
Other: Physiotherapy ASPETAR — Standardized physiotherapy protocol
  Arms: Physiotherapy ASPETAR
Other: Physiotherapy ASPETAR+ — Standardized physiotherapy protocol including early lengthening exercises
  Arms: Physiotherapy ASPETAR+

SUMMARY:
The purpose of the study is to compare the effect of two rehabilitation protocols with different emphasis on eccentric exercises after acute hamstring muscle strain injuries on the time to return to sports (RTS) and the rate of re-injuries in male athletes.

The hypothesis is that the addition of early eccentric hamstring exercises being performed at longer muscle-tendon length towards end range of motion alter the outcomes RTS and re-injuries in a rehabilitation protocol after acute hamstring muscle strain injuries.

DETAILED DESCRIPTION:
Background and rationale:

Acute hamstring muscle strain injuries represent the most prevalent non-contact muscle injury reported in sports. Despite the high prevalence and a rapidly expanding body of literature investigating hamstring muscle strain injuries, [1] occurrence and re-injury rates have not improved over the last three decades [2]. Therefore, rehabilitation and secondary prevention are of particular concern, and the primary objective of all rehabilitation protocols is to return an athlete to pre-injury level as soon as possible with a minimal risk of injury recurrence.There is still a lack of consensus and clinical research regarding the effectiveness of various rehabilitation protocols for acute hamstring injuries in athletes participating in sports with high sprinting demands [3,4]. To our knowledge, there are no prospective, randomised trials investigating the effect of different rehabilitation protocols in a Middle-Eastern athletic population. Eccentric strength training has shown to reduce the risk of both new acute hamstring injuries as well as re-injuries [5,6], whereas hamstring exercises being performed at longer muscle-tendon length, preferentially mimicking movements occuring simultaneously at both the knee and hip are reported to be more effective than a protocol containing conventional exercises [7], and are suggested to be a key strategy in the management of hamstring injuries. However, the preventive effect related to the eccentric training remains unclear and is still debated and the optimal intensity of eccentric training in rehabilitation of acute hamstring strain injuries and prevention of re-injuries is yet unknown [8].

The primary objective in this study is therefore to compare the effect of two rehabilitation protocols after acute hamstring muscle strain injuries on the time to return to sports (RTS) and the rate of re-injuries in male athletes in a prospective single-site randomized controlled trial.

The investigators aim to include 90 male athletes with clinical signs and MRI abnormalities consistent with an acute hamstring muscle strain injury. The injured athletes will be randomised into one of two different rehabilitation protocols with unlike emphasis on eccentric exercises.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes
* Age 18-50 years
* Acute onset posterior thigh pain when training or competing, identified as:

  1. Patient reported sudden event
  2. Patient reported pain in posterior thigh
* Clinical diagnosis of an acute hamstring muscle strain injury, defined as:

  1. Localised pain during palpation of hamstring muscle
  2. Increasing pain during isometric contraction
  3. Localised pain when performing a passive straight leg raise test
* MRI confirmed isolated hamstring lesion (increased high signal intensity on fat saturated sequences)
* MRI performed ≤5 days from injury
* Available for ≥3 physiotherapy sessions per week at Aspetar
* Available for follow-up

Exclusion Criteria:

* Patients with verified or suspected previous hamstring injury within the last 6 months in the same leg
* Chronic hamstring complaints >2 months
* Grade III injury including complete hamstring disruption or avulsion of all tendons
* Contraindications to MRI
* Patients that do not have an intention to return to full sport activity
* Patients that do not want to receive one of the two therapies

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-03; Primary Completion 2019-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Time to Return to Sport (RTS) | After the initial injury, patients will be followed daily during working days for the duration of time until they return to RTS, with an expected average of 25 days up to 1 year
  Number of days between initial injury and return to full unrestricted training and/or match play

SECONDARY OUTCOMES:
Re-injury within 2 months, 6 months and 12 months after RTS | The patients will be monitored by phone 2 months, 6 months and 12 months after RTS
  In the event of a clinical suspicion of re-injury, the player will be advised to immediately call the primary investigator and consult a physician

OTHER OUTCOMES:
Subjective pain score assessed with visual analogue scale (VAS) | Measured initial at inclusion, daily up to 5 days a week throughout the rehabilitation period and at RTS with an expected average of 25 days up to 1 year
  pain evaluation
Pain during walking and jogging | Measured initial at inclusion, daily up to 5 days a week throughout the rehabilitation period and at RTS with an expected average of 25 days up to 1 year
  pain evaluation
Pain and restriction during with trunk flexion | Measured initial at inclusion, daily up to 5 days a week throughout the rehabilitation period and at RTS with an expected average of 25 days up to 1 year
  pain evaluation
Length and width of painful area with palpation | Measured initial at inclusion, daily up to 5 days a week throughout the rehabilitation period and at RTSwith an expected average of 25 days up to 1 year
  palpation evaluation
Distance from tuber to maximal painful area identified with palpation | Measured initial at inclusion and at RTS with an expected average of 25 days up to 1 year
  palpation evaluation
Hamstring force | Mid range, outer range measured initial at inclusion, daily up to 5 days/w throughout the rehab. period and at RTS with expected average 25 days - up to 1 year. Inner range measured at initial inclusion and RTS with expected 25 days up to 1 year
  Inner range, mid range and outer range hamstring force measured with handheld dynamometry (HHD) [9]
Hamstring flexibility | SLR and MHFAKE measured initial at inclusion, daily up to 5 days a week throughout the rehabilitation period and at RTS with expected average 25 days up to 1 year. PKET measured initial at inclusion and at RTS with expected average 25 days up to 1 year
  Hamstring flexibility measured as passive straight leg raise (SLR), passive knee extension (PKET) and maximal hip flexion active knee extension (MHFAKE) with inclinometer
Painful single leg bridge | Measured initial at inclusion, daily up to 5 days a week throughout the rehabilitation period and at RTS with an expected average of 25 days up to 1 year
  functional pain evaluation
Patient prediction | Measured initial at inclusion
  Patient prediction on time to RTS and performance after RTS
MRI parameters | Measured initial at inclusion
  MRI evaluation
Isokinetic knee flexor strength | Measured initial (uninjured leg) at inclusion and at RTS (both legs) with an expected average of 25 days up to 1 year
  Isokinetic knee flexor strength assessed with BIODEX
Eccentric knee flexor strength during Nordic Hamstring Exercise | Measured at RTS with an expected average of 25 days up to 1 year
  Eccentric knee flexor strength measured during Nordic Hamstring Exercise performed on a Novel Device
sEMG hamstring muscle activity | Measured initial at inclusion and at RTS with an expected average of 25 days up to 1 year
  sEMG is measured during isokinetic knee flexor strength testing with BIODEX initial on uninjured leg and at RTS on both legs. sEMG is measured during eccentric knee flexor strength test performed (Nordic Hamstring Exercise) at RTS.
Insecurity with dynamic flexibility test (H-test) [10] | Measured at RTS with an expected average of 25 days up to 1 year
  Htest evaluation
RTS questions | Measured at RTS with an expected average of 25 days up to 1 year
  RTS questions including rate of recovery and fear of sustaining a new injury
Days between injury and 1st training with the club team and 1st match played | The patients are monitored by phone after RTS with an expected average of 25 days up to 1 year
  evalaution number of days training

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Whiteley, PhD, PT, Principal Investigator — Aspetar Orthopaedic and Sports Medicine Hospital; Arnlaug Wangensteen, MSc, Study Director — Aspetar Orthopaedic and Sports Medicine Hospital, Norwegian School for Sports Science; Roald Bahr, Prof. PhD MD, Study Director — Aspetar Orthopaedic and Sports Medicine Hospital; Erik Witvrouw, Prof. PhD PT, Study Director — Aspetar Orthopaedic and Sports Medicine Hoslpital; Johannes Tol, PhD MD, Study Director — Aspetar Orthopaedic and Sports Medicine Hospital
Locations (1):
- Aspetar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamilton B. Hamstring muscle strain injuries: what can we learn from history? Br J Sports Med. 2012 Oct;46(13):900-3. doi: 10.1136/bjsports-2012-090931. Epub 2012 Mar 29. No abstract available. PMID 22460740
- [Background] Kerkhoffs GM, van Es N, Wieldraaijer T, Sierevelt IN, Ekstrand J, van Dijk CN. Diagnosis and prognosis of acute hamstring injuries in athletes. Knee Surg Sports Traumatol Arthrosc. 2013 Feb;21(2):500-9. doi: 10.1007/s00167-012-2055-x. Epub 2012 May 24. PMID 22622781
- [Background] Reurink G, Goudswaard GJ, Tol JL, Verhaar JA, Weir A, Moen MH. Therapeutic interventions for acute hamstring injuries: a systematic review. Br J Sports Med. 2012 Feb;46(2):103-9. doi: 10.1136/bjsports-2011-090447. Epub 2011 Oct 28. PMID 22039218
- [Background] Mason DL, Dickens VA, Vail A. Rehabilitation for hamstring injuries. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004575. doi: 10.1002/14651858.CD004575.pub3. PMID 23235611
- [Background] Arnason A, Andersen TE, Holme I, Engebretsen L, Bahr R. Prevention of hamstring strains in elite soccer: an intervention study. Scand J Med Sci Sports. 2008 Feb;18(1):40-8. doi: 10.1111/j.1600-0838.2006.00634.x. Epub 2007 Mar 12. PMID 17355322
- [Background] Petersen J, Thorborg K, Nielsen MB, Budtz-Jorgensen E, Holmich P. Preventive effect of eccentric training on acute hamstring injuries in men's soccer: a cluster-randomized controlled trial. Am J Sports Med. 2011 Nov;39(11):2296-303. doi: 10.1177/0363546511419277. Epub 2011 Aug 8. PMID 21825112
- [Background] Askling CM, Tengvar M, Thorstensson A. Acute hamstring injuries in Swedish elite football: a prospective randomised controlled clinical trial comparing two rehabilitation protocols. Br J Sports Med. 2013 Oct;47(15):953-9. doi: 10.1136/bjsports-2013-092165. Epub 2013 Mar 27. PMID 23536466
- [Background] Malliaropoulos N, Mendiguchia J, Pehlivanidis H, Papadopoulou S, Valle X, Malliaras P, Maffulli N. Hamstring exercises for track and field athletes: injury and exercise biomechanics, and possible implications for exercise selection and primary prevention. Br J Sports Med. 2012 Sep;46(12):846-51. doi: 10.1136/bjsports-2011-090474. Epub 2012 Jun 9. PMID 22685125
- [Background] Whiteley R, Jacobsen P, Prior S, Skazalski C, Otten R, Johnson A. Correlation of isokinetic and novel hand-held dynamometry measures of knee flexion and extension strength testing. J Sci Med Sport. 2012 Sep;15(5):444-50. doi: 10.1016/j.jsams.2012.01.003. Epub 2012 Mar 15. PMID 22424705
- [Background] Askling CM, Nilsson J, Thorstensson A. A new hamstring test to complement the common clinical examination before return to sport after injury. Knee Surg Sports Traumatol Arthrosc. 2010 Dec;18(12):1798-803. doi: 10.1007/s00167-010-1265-3. Epub 2010 Sep 18. PMID 20852842
- [Background] Tol JL, Hamilton B, Eirale C, Muxart P, Jacobsen P, Whiteley R. At return to play following hamstring injury the majority of professional football players have residual isokinetic deficits. Br J Sports Med. 2014 Sep;48(18):1364-9. doi: 10.1136/bjsports-2013-093016. Epub 2014 Feb 3. PMID 24493666
- [Derived] Zein MI, Mokkenstorm MJK, Cardinale M, Holtzhausen L, Whiteley R, Moen MH, Reurink G, Tol JL; Qatari and Dutch Hamstring Study Group. Baseline clinical and MRI risk factors for hamstring reinjury showing the value of performing baseline MRI and delaying return to play: a multicentre, prospective cohort of 330 acute hamstring injuries. Br J Sports Med. 2024 Jul 1;58(14):766-776. doi: 10.1136/bjsports-2023-107878. PMID 38729628
- [Derived] Whiteley R, van Dyk N, Wangensteen A, Hansen C. Clinical implications from daily physiotherapy examination of 131 acute hamstring injuries and their association with running speed and rehabilitation progression. Br J Sports Med. 2018 Mar;52(5):303-310. doi: 10.1136/bjsports-2017-097616. Epub 2017 Oct 30. PMID 29084725